CLINICAL TRIAL: NCT02184663
Title: Multicenter, Randomized Study, Evaluation of Adapted Physical Activity Program in Patients With Unresectable, Locally Advanced or Metastatic Pancreatic Cancer
Brief Title: Evaluation of an Adapted Physical Activity Program in Patients With Unresectable Pancreatic Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: APACaP D13-1; 2014-A00228-39 (Other: ANSM)
Record Dates: First submitted 2014-07-02; First posted 2014-07-09 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Unresectable Locally Advanced Cancer; Metastatic Pancreatic Cancer
Keywords: Unresectable; Pancreatic cancer; GERCOR; Adapted physical activity (APA); Quality of life; Fatigue
MeSH Terms: conditions — Pancreatic Neoplasms; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care without APA program (Active Comparator): The control arm corresponds to usual care (without APA), including :
  * Weekday hospital chemotherapy (every 7 or 14 days, depending on chemotherapy protocol)
  * Evaluation by the oncologist at the usual rate
  * Assessment every 8 weeks (TAP scan + CA-19.9)
  * Nutritional, psychological and pain management as recommended, according to the usual schedule.
  Interventions: Other: without APA program
- Standard care with APA program (Experimental): The experimental arm corresponds to usual care, combined with a 16-week APA program.
  The APA program consisted of personalized aerobic and resistance exercises, with a weekly remote supervision by an APA professional trainer, and unsupervised sessions with a family member or friend (APA partner).
  Interventions: Other: APA program

INTERVENTIONS:
Other: without APA program — Control Arm : chemotherapy alone
  Arms: Standard care without APA program
Other: APA program — Experimental Arm : chemotherapy + APA program during 16 weeks (aerobic and muscular strength exercises)
  Arms: Standard care with APA program

SUMMARY:
Adapted Physical Activity (APA) program may provide an opportunity to improve symptoms for patients with unresectable pancreatic cancer.

Thereby, it is proposed to conduct an open trial to assess effects of the APA program in such population

DETAILED DESCRIPTION:
The benefit of Adapted Physical Activity (APA) has been demonstrated after cancer diagnosis in term of symptomatic improvement: reducing fatigue, pain and improving the quality of life, psychological and emotional state, and adherence to treatment.

The aim of the study is to assess the effects of an APA program in pancreatic cancer population treated by usual chemotherapy.

200 randomized patients are required.

The program is organized in 16 weeks. During the trial, assessments include: aerobic exercises, muscular strength, six-minute walk test, body composition (bioimpedance, L3 CT-scan), level of physical activity - International Physical Activity Questionnaire - (IPAQ questionnaire), fatigue - Multidimensional Fatigue Inventory - (MFI-20 questionnaire), quality of life - EORTC Quality of Life questionnaire C-30 - (EORTC QLQ-30 questionnaire), depression symptom - Hospital Anxiety and depression scale - (HADS questionnaire), pain (Brief Pain Inventory Short form), and nutritional evaluation (BMI, ingests EVA).

Furthermore, relationships between insulin resistance, insulin secretion, Insulin like Growth Factor 1 (IGF-1) and pancreatic carcinogenesis exist. APA may improve the quality of life in decreasing insulin-resistance, insulin secretion and IGF-1.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven non resectable pancreatic adenocarcinoma
* Indication of palliative chemotherapy
* Life expectancy ≥ 3 months
* Eastern Cooperative oncology group (ECOG) - Performance status ≤2
* Age ≥18 years old
* At least one measurable lesion as assessed by CT-scan or MRI (Magnetic resonance Imaging)
* Identified Accompanying partner Adapted Physical Activity (AAPA)
* Signed and dated informed consent
* Registration in a National Health Care System (CMU included for France)

Exclusion Criteria:

* Previous Cerebrovascular accident or myocardial infarction <6months
* Uncontrolled hypertension.
* Severe cardiovascular or respiratory disease
* Severe cognitive or psychiatric disorder
* Severe motor and/or sensory neuropathy
* Rheumatologic or orthopedic problem or bone lesions with a fracture risk
* Others comorbidities contra-indicated physical exercises
* Patient protected by the law - Guardianship and trusteeship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2014-11-20 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life (HRQoL) at 16 weeks | At 16 weeks
  HRQoL at week 16 according to the EORTC Core Quality of Life questionnaire (EORTC QLQ-C30) with three targeted dimensions: global health status, physical function and fatigue.

SECONDARY OUTCOMES:
Time To deterioration (TTD) | Up to 24 months
Brief Pain Inventory Short form questionnaire | Up to 24 months
Patient depression scale - HADS questionnaire | Up to 24 months
Nutritional status evaluation | up to 24 months
  Nutritional Status will be measured by weigth, Body Mass Index, body composition, EVA ingests, caloric intake and protidic, albumin/prealbumin, inflammation markers (PNN and CRP)
Physical Activity evaluation - IPAQ questionnaire | up to 24 months
  Six minutes walk test, dyspnea scale, Borg scale, muscular pain, strength test with bands and compliance program
Number of Adverse events (AE) grade 3 -4 | up to 24 months
Progression free survival (PFS) | 2 years
Overall Survival (OS) | 2 years
Accompanying partner depression scale (HADS questionnaire) | up to 24 months
General state - Performance status OMS | up to 24 months
Fatigue scale (EVA fatigue) | up to 24 months
MFI-20 and EORTC QLQ C-30 evaluation | at 6, 12 et 24 months
medico-economic evaluation | up to 24 months
visual analog scale for pain | up to 24 months
analgesic consumption | up to 24 months
anxiolytic / antidepressant consumption | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Hammel, MD, Principal Investigator — Hôpital Beaujon
Locations (17):
- France (17):
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - CHU Morvan, Brest
  - Hôpital Beaujon, Clichy
  - Hôpital Henri Mondor, Créteil
  - Centre Georges François Leclerc, Dijon
  - CHD Vendée, La Roche-sur-Yon
  - Institut Hospitalier Franco-Britannique, Levallois-Perret
  - Centre Léon Bérard, Lyon
  - CH Saint Joseph Saint Luc, Lyon
  - Hôpital Européen, Marseille
  - CH Mont de Marsan, Mont-de-Marsan
  - Centre Hospitalier de Belfort, Montbéliard
  - Hôpital Cochin, Paris
  - Hôpital Saint Antoine, Paris
  - CHU Robert Debré, Reims
  - Hôpital FOCH, Suresnes
  - Institut de cancérologie de Lorraine, Vandœuvre-lès-Nancy

REFERENCES:
- [Derived] Neuzillet C, Vergnault M, Bonnetain F, Hammel P. Rationale and design of the Adapted Physical Activity in advanced Pancreatic Cancer patients (APACaP) GERCOR (Groupe Cooperateur Multidisciplinaire en Oncologie) trial: study protocol for a randomized controlled trial. Trials. 2015 Oct 12;16:454. doi: 10.1186/s13063-015-0983-8. PMID 26458923